CLINICAL TRIAL: NCT05657054
Title: Effect of an Exercise Intervention Targeting Hip Strengthening in Patients Undergoing Revision Total Hip Replacement - a Multicenter, Randomized Controlled Trial (The Strong Hip Trial)
Brief Title: Exercise Intervention Targeting Hip Strengthening Compared to Usual Care in Patients Undergoing Revision Hip Replacement
Acronym: StrongHip
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Vejle Hospital (Other); Regionshospitalet Silkeborg (Other); Gødstrup Hospital (Other); Viborg Regional Hospital (Other); Odense University Hospital (Other); Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StrongHip
Record Dates: First submitted 2022-11-24; First posted 2022-12-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Revision Total Hip Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength group (Experimental): Group 1
  Interventions: Other: Exercise Intervention Targeting Hip Strengthening
- Control group (Active Comparator): Group 2
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Exercise Intervention Targeting Hip Strengthening — An initial 16-week exercise intervention of 45 minutes of training 3 times a week in the patient's own home or at a rehabilitation center. Patients will be instructed by a physiotherapist during the first 3 sessions, in order to be able to perform the exercises at home. Subsequently, there are physiotherapist-supervised sessions once every second week. The delivery of the supervised sessions is based on the patient's preferences, either by physical attendance or remotely in the patient's home. The intervention will consist of 4 exercises adapted from the NEMEX program targeting lower extremity muscle strength, stability, postural function, and postural orientation. Progression is made when an exercise is performed with good sensorimotor control and good performance quality and with minimal exertion and adequate movement control. Progression is primarily provided by 3 levels of difficulty and secondly by varying the number of repetitions or where possible, by increasing the weight load.
  Arms: Strength group
Other: Usual Care — The intervention will consist of a rehabilitation intervention corresponding to standard care in the participating municipalities (i.e. content and duration of intervention). The intervention will be delivered individually or as group training, based on a clinical assessment of the individual patients' needs. The intervention can be supported by home-based exercises following instruction from a physiotherapist, supplemented by the provision of written information or access to a virtual training program. The intervention occurs in either the rehabilitation center's gym or the patient's home. The training sessions may consist of some of the following parameters: Strength training, stretching, functional training e.g. walking and stair climbing, stability training, balance training, endurance training, and gait correction.
  Arms: Control group

SUMMARY:
There is sparse evidence on revision total hip replacement (THR), regarding the effectiveness on pain and function, and no consensus exists on optimal rehabilitation after revision THR. Further, patients undergoing revision THR achieve worse clinical outcomes on hip pain and function compared to patients undergoing primary THR. The primary aim of this randomized controlled trial is to compare the clinical effectiveness of a partly tele-delivered exercise intervention targeting hip strengthening with the standard community-based rehabilitation (usual care) in patients undergoing revision THR. The investigators will test the hypothesis that the exercise intervention targeting hip strengthening is superior to standard community-based rehabilitation in improving physical function measured with the 30-second Chair Stand Test at 16-week follow-up.

DETAILED DESCRIPTION:
There is sparse evidence on revision total hip replacement (THR), regarding the effectiveness on pain and function, and no consensus exists on optimal rehabilitation after revision THR. Revision THR is one of the more technically challenging orthopedic surgeries and patients undergoing revision THR report improvements in pain and function. Nevertheless, patients undergoing revision THR achieve worse clinical outcomes on hip pain and function compared to patients undergoing primary THR. This calls for research exploring different rehabilitation approaches, in order to improve clinical outcomes for patients after revision THR.

This study aims to compare the clinical effectiveness of a partly tele-delivered exercise intervention targeting hip strengthening with the standard community-based rehabilitation (usual care) in patients undergoing revision THR.

This randomized, controlled, assessor-blinded trial is a multicenter trial involving hospitals and municipality rehabilitation centers across Denmark. Eligible patients undergoing revision THR will be randomized into two groups: A partly remotely-delivered hip strengthening rehabilitation intervention (strength group) or usual care (control group).

The exercise intervention targeting hip strengthening will partly follow the Neuromuscular Exercise (NEMEX) program as described by Eva Ageberg et al., and the intervention is further modified based on expert opinion from patients' experience with rehabilitation from a prior qualitative study. Usual care consists of rehabilitation in the municipalities, where it is up to the individual physiotherapist and the municipality to organize the rehabilitation, which is why both type, content, and duration may vary.

The primary outcome will be change in functional performance measured by the 30-second Chair Stand Test. Outcomes will be measured at baseline, after 16 weeks of intervention, and at 12-month follow-up.

The investigators hypothesize that the exercise intervention targeting hip strengthening is superior to usual care in improving physical function measured with the 30-second Chair Stand Test at 16-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first revision THR
* Age ≥ 18 years
* Motivated to participate in an exercise program for 16 weeks
* Provided informed consent to participate
* Patients who has the cup and/or stem replaced or a combination of liner and caput replaced
* Patients who can be baseline tested (chair stand test, stair climb test, 40m walking test)

Exclusion Criteria:

* Dependency of wheelchair
* Preplanned other lower limb surgery within 12 months
* Body Mass Index (BMI) score > 40
* Currently undergoing cancer treatment, e.g. chemo-, immuno-, or radiotherapy.
* Comorbidities that prevent exercise
* Inadequacy in written and spoken Danish
* Mentally unable to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in functional performance measured by the 30-seconds chair stand test | Measured at baseline, 16-week, and 12-month follow-up.
  The 30-second chair stand test is a valid and reliable measure of lower-extremity muscle strength evaluating sit-to-stand function, which is limited in people undergoing hip replacement.

SECONDARY OUTCOMES:
Change in the Hip disability and Osteoarthritis Outcome Score (HOOS) pain subscale | Measured at baseline, 16-week, and 12-month follow-up.
  The HOOS pain subscale is a 10-item patient-reported outcome measure designed to assess hip pain in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better pain status.
Change in the HOOS symptoms subscale | Measured at baseline, 16-week, and 12-month follow-up.
  The HOOS symptom subscale is a five-item patient-reported outcome measure designed to assess other hip symptoms in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better symptom status.
Change in the HOOS activities of daily living (ADL) function subscale | Measured at baseline, 16-week, and 12-month follow-up.
  The HOOS ADL function subscale is a 17-item patient-reported outcome measure designed to assess ADL function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better ADL function status.
Change in the HOOS quality-of-life subscale | Measured at baseline, 16-week, and 12-month follow-up.
  The HOOS quality-of-life subscale is a four-item patient-reported outcome measure designed to assess hip-related quality-of-life in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better quality-of-life status.
Change in the HOOS sports and recreation subscale | Measured at baseline, 16-week, and 12-month follow-up.
  The HOOS sports and recreation subscale is a four-item patient-reported outcome measure designed to assess sports and recreation function in patients with hip osteoarthritis. The total score ranges from 0 to 100, with higher scores indicating better sports and recreation status.
Change in 40m Fast-Paced Walk Test (40m-FPWT) | Measured at baseline, 16-week, and 12-month follow-up.
  The 40m-FPWT is a physical function test designed to measure the ability to walk quickly over short distances and is measured as the time it takes to complete a 40 m course at a fast walking pace.
Change in 9-step Timed Stair Climb Test (9-step TSCT) | Measured at baseline, 16-week, and 12-month follow-up.
  The 9-step TSCT is a physical function test designed to measure lower body strength and balance as well as ascending and descending stair activity and is measured as the time it takes to ascend and descend a 9-step stair.
Change in leg extension muscle power (watt/kg body weight) | Measured at baseline, 16-week, and 12-month follow-up.
  The Nottingham Power Rig (NPR) is used to measure leg extensor muscle power. The NPR measures the power output in total watt and watt pr. bodyweight in kilograms from a seated push on a flat pedal which is transmitted by a lever and chain to spin a flywheel. The NPR is a safe and reliable method to measure explosive knee extensor muscle power and has been validated as a clinically important measure of muscle function in elderly individuals.
Global Perceived Effect (GPE) | Measured at 16-week and 12-month follow-up.
  The GPE will be used as a measure of patient-rated recovery and will be assessed for three domains; pain, activities of daily living, and quality of life rated on a 7-point Likert scale ranging from 'very bad' (worst) to 'very good' (best)
AE (Adverse Events) & Serious Adverse Events (SAE) | Registered throughout the 12-month study period.
  Continuous registration of health issues and injuries. The events will be monitored by the physiotherapists supervising the exercise sessions. Further, patients will be asked at 4- and 12-month follow-ups about potential AE and SAE using open-probe questions.
Adherence to the 16-week intervention | Registered throughout the 16-week initial intervention.
  High adherence is defined as attendance in ≥75% of the exercise sessions.
Drop-outs | Registered throughout the 12-month study period.
  Number of drop-out from the interventions.

OTHER OUTCOMES:
Physical activity | Measured at 12-week and 12-month follow-up.
  Physical activity will be measured by The International Physical Activity Questionnaires (IPAQ), which is a 7 items questionnaire consisting of open-ended questions surrounding the patient's last 7-day recall of physical activity.
Change in pain measured on a Numerical Rating Scale (NRS) | Measured at baseline, 16-week, and 12-month follow-up.
  NRS pain score will be measured before and after each exercise session and at each follow-up evaluation before completing the functional performance tests. The 11-point numeric scale ranges from '0' representing "no pain" (best) to '10' representing "worst pain imaginable" (worst).
Change in EuroQol Group 5-Dimension 5-Level (EQ-5D-5L) | Measured at baseline, 16-week, and 12-month follow-up.
  The EQ-5D-5L is a five-item patient-reported outcome measure designed to assess generic health-related quality of life. The total score of the descriptive index and EuroQol Visual Analogue Scale (EQ-VAS) ranges from -0.624 (worst) to 1.000 (best) and 0 (worst imaginable health) to 100 (best imaginable health), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Stisen, MSc, Principal Investigator — Aarhus University Hospital and Aarhus University; Inger Mechlenburg, Prof., Study Director — Aarhus University Hospital and Aarhus University; Alma B Pedersen, Prof., Study Director — Aarhus University Hospital and Aarhus University; Troels Kjeldsen, MSc, Study Director — Aarhus University Hospital and Aarhus University
Locations (9):
- Denmark (9):
  - Aarhus University, Aarhus
  - Aarhus University Hospital, Aarhus N
  - Bispebjerg Hospital, Copenhagen
  - University Hospital, Gentofte, Copenhagen, Hellerup
  - Gødstrup Hospital, Herning
  - Odense University Hospital, Odense
  - Regional Hospital Silkeborg, Silkeborg
  - Vejle Hospital, Vejle
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Yes
Anonymised patient-level data for the primary and all secondary outcome measures will be made available if required by the scientific journal, in which the results of the trial are published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after publication of the trial.
Access Criteria: Data access will be reviewed by the author group. Requesters will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Stisen MG, Pedersen AB, Kjeldsen T, Foldager FN, Lamm M, Assenholt A, Hvidberg KL, Rasmussen MK, Aalund PK, Frandsen CF, Holsgaard-Larsen A, Haubro MH, Bieler T, Overgaard S, Beck T, Ingwersen KG, Parner ET, Mechlenburg I. Hip strengthening exercise compared to standard rehabilitation after revision hip replacement: a multicenter randomized controlled trial. Ann Phys Rehabil Med. 2026 Jan 13;69(4):102076. doi: 10.1016/j.rehab.2025.102076. Online ahead of print. PMID 41534141
- [Derived] Stisen MB, Pedersen AB, Kjeldsen T, Mechlenburg I. Effect of an exercise intervention targeting hip strengthening in patients undergoing revision total hip replacement-A study protocol for a multicenter randomized controlled trial. Physiother Res Int. 2024 Jul;29(3):e2101. doi: 10.1002/pri.2101. PMID 38859640

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT05657054/SAP_000.pdf